CLINICAL TRIAL: NCT05817786
Title: Treatment of Upper Limb Chronic Neuropathic Pain by Electrical Stimulation of the Brachial Plexus Nerve Roots
Acronym: SIMPLEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-APN-01; 2021-A02538-33 (Other: ANSM)
Record Dates: First submitted 2023-03-31; First posted 2023-04-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: randomisation at month 1
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BP PNS (experimental group) (Experimental): Patients with refractory upper limb neuropathic pain treated by chronic electrical stimulation of the brachial plexus nerve roots
  Interventions: Device: electrical stimulation of the brachial plexus nerve roots
- sham stimulation (control group). (Active Comparator): Patients with refractory upper limb neuropathic pain treated by sham stimulation
  Interventions: Other: sham stimulation

INTERVENTIONS:
Device: electrical stimulation of the brachial plexus nerve roots — treated by chronic electrical stimulation of the brachial plexus nerve roots
  Arms: BP PNS (experimental group)
Other: sham stimulation — treated by sham stimulation
  Arms: sham stimulation (control group).

SUMMARY:
Moderate to severe neuropathic pain has a prevalence of 5% in the French population, involving the upper limb (UL) in 47%. Invasive neuromodulation, mainly spinal cord stimulation (SCS) is recommended as a third line treatment in refractory chronic neuropathic pain when optimized medical treatments are not sufficient to control pain.

The implantation technique for BP roots PNS is based on the ultrasound-guided percutaneous inter-scalenic approach, routinely used for BP anesthetic blocks. As for SCS, BP PNS relies on chronic electrical stimulation of the nerve roots via chronically implanted devices (one lead connected to a subcutaneous generator).

However efficacy of BP PNS has never been evaluated in controlled conditions. Our objectives are to assess, in controlled conditions, the effects of BP PNS in term of pain relief, quality of life improvement and safety.

DETAILED DESCRIPTION:
Moderate to severe neuropathic pain has a prevalence of 5% in the French population, involving the upper limb (UL) in 47% . Invasive neuromodulation, mainly spinal cord stimulation (SCS) is recommended as a third line treatment in refractory chronic neuropathic pain when optimized medical treatments are not sufficient to control pain. However, SCS implanted at the cervical level, required to control UL pain, has shown its efficacy but has specific technical issues that limit its use: lead dislocation or breakage (0-43%), lead migration (0-12,5%), unwanted paresthesias in the trunk or the lower limb(s) (17%), paresthesias changes during head movements (48%). To avoid these limitations, peripheral nerve stimulation (PNS) targeting the UL nerve trunks or nerve roots of the brachial plexus (BP) has been proposed in short pioneering series reporting encouraging results .

The implantation technique for BP roots PNS is based on the ultrasound-guided percutaneous inter-scalenic approach, routinely used for BP anesthetic blocks. As for SCS, BP PNS relies on chronic electrical stimulation of the nerve roots via chronically implanted devices (one lead connected to a subcutaneous generator).

In a recent prospective series of 26 patients suffering from UL refractory pain, we reported that 20 patients still using the stimulation at last follow-up (28 months) experienced a mean pain relief of 67%. Seventeen patients were improved ≥50%, including 12 improved ≥70%. Complications were rare: stimulation intolerance due to shock-like sensations, superficial infection, lead fractures and lead migration . However efficacy of BP PNS has never been evaluated in controlled conditions. Our objectives are to assess, in controlled conditions, the effects of BP PNS in term of pain relief, quality of life improvement and safety.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility will be determined by trained clinicians with expertise in chronic pain and neuropathic pain.
* Patients between 18 and 80 years old
* suffering from moderate to severe (VAS score >5/10) chronic (duration> 12 months) neuropathic (DN4 score ≥ 4/10) unilateral pain - located in the upper limb.
* from peripheral origin, including complex regional pain syndrome type I and II, post-traumatic or post surgical pain.
* refractory to first and second line treatments for neuropathic pain according recent French recommendations and guidelines[6], including serotonin- noradrenaline reuptake inhibitor (SNRI) antidepressants (duloxetine and venlafaxine), gabapentin, pregabalin, tricyclic antidepressants, topical lidocaine, high-concentration capsaicin patches, psychotherapy and combinations of them.

Patient have signed informed consent

- Patient benefiting from French social insurance system

Exclusion Criteria:

* Brachial plexus avulsion
* Post-zoster neuropathic pain
* Phantom limb pain
* Patient unable to fill a self-administered questionnaire
* Patients with a chronic disease requiring repeated MRI monitoring
* Patients with contra-indication to general anesthesia, surgery or percutaneous BP approach.
* Patients with other pacemakers (cardiac pacemaker or defibrillator) or patients with a high risk to use a defibrillator due to a known cardiac disorder.
* Patients with instable neuropsychological or psychiatric disorders
* Vulnerable patients: pregnant or breast feeding, minor, adult under guardianship or deprived freedom

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
efficacity | after 3 months of treatment
  evaluation by the patient with quizz EQ5D (worse: 0-better: 20)
efficacity | after 3 months of treatment
  evaluation by the patient with quizz VAS (worse: 0- better: 100)

CONTACTS AND LOCATIONS:
Overall Officials: Denys FONTAINE, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - CHU de Lyon, Lyon, France
  - CHU de Nice, Nice, France
  - CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No